CLINICAL TRIAL: NCT01791881
Title: Double-blinded, Randomized, Active Control Comparative, Parallel-designed, Phase III Clinical Trial: Therapeutic Confirmatory Clinical Trial to Evaluate the Safety and Efficacy of "Hugeltox Inj." In Essential Blepharospasm Running Parallel With Phase I Study
Brief Title: Therapeutic Confirmatory Clinical Trial to Evaluate the Safety and Efficacy of "Hugeltox Inj." in Essential Blepharospasm
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hugel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HG-06-01
Record Dates: First submitted 2013-02-13; First posted 2013-02-15 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Essential Blepharospasm
MeSH Terms: conditions — Benign essential blepharospasm | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Botulinum toxin type A(Botox®) (Active Comparator): Botulinum toxin type A(Botox®)
  Interventions: Drug: Hugeltox; Drug: Botulinum Toxin Type A(Botox®)
- Botulinum toxin type A(Hugeltox) (Experimental): Botulinum toxin type A(Hugeltox)
  Interventions: Drug: Hugeltox; Drug: Botulinum Toxin Type A(Botox®)

INTERVENTIONS:
Drug: Hugeltox — 1.25U~2.5U/site, Maximum dosage 12.5U~60U/person
Drug: Botulinum Toxin Type A(Botox®) — 1.25U~2.5U/site, Maximum dosage 12.5U~60U/person

SUMMARY:
To compare the efficacy and safety of Hugel-Tox (Botulinum toxin A, Hugel, Korea) against Botox in the treatment of Essential Blepharospasm and to get a regulatory approval from KFDA

ELIGIBILITY:
Inclusion Criteria:

* Adult between ages 18 and 75 years
* All patients, diagnosed of essential blepharospasm, with Grade 2~4 of Severity of Spmasm (by Scott's Method)

Exclusion Criteria:

* Patients have undergone surgical surgery to treat blepharospmasm like myectomy or neurectomy
* Patients with hypersensitivity history to botulinum toxin products previously
* Patients with secondary blepharomspasm
* Patients with hemifacialspasm
* Patients with treatment following drugs ; Anticonvulsants, tranquilizers, narcotics, aminoglycoside antibiotics, muscle relaxtants like baclofen etc., blockers of parasympathetic nervous system, levodopa
* Patients with previous injection of other botulinum toxin products in 3 months
* Patients with any other significant neuromuscular disease like Myasthenia gravis
* Pregnant or breastfeeding women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2008-04; Primary Completion 2009-05 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Rate of patients with an improvement more than one Grade of Severity of Spasm (by Scott's Method) | at 4 weeks post-injection

SECONDARY OUTCOMES:
(1) Duration of action days | 6 months
(2) Grades of Severity of Spasm (by Scott's Method), Functional Visual Status | at four weeks post-injection
(3) Rate of patients with a Grade-0 or Grade-1 of Severity Spasm (by Scott's Method) | at four weeks post-injection
(4) Rate of patients with an improvement more than two Grade of Severity of Spasm (by Scott's Method) | at four weeks post-injection

CONTACTS AND LOCATIONS:
Overall Officials: Yoon-Duck Kim, M.D., Ph.D., Study Chair — Samsung Medical Center
Locations (9):
- South Korea (9):
  - Samsung medical Center, Seoul, Seoul
  - The Catholic University, Seoul, St.Mary's hospital, Seoul, Seoul
  - Cha Hospital, Bundang
  - Seoul National University Hospital - Bundang, Bundang
  - Youngnam University Hospital, Daegu
  - Chungang University Hospital, Seoul
  - Kim's eye hospital, Seoul
  - The catholic university, Yeouido, St. Mary's hospital, Seoul
  - Yeonsei University, Severance hospital - Gangnam, Seoul